CLINICAL TRIAL: NCT00194987
Title: A Randomized Multicenter Trial of Antenatal Treatment of Alloimmune Thrombocytopenia
Brief Title: A Trial of Antenatal Treatment of Alloimmune Thrombocytopenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0102004801
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Alloimmune Thrombocytopenia; Fetal Alloimmune Thrombocytopenia
Keywords: Alloimmune thrombocytopenia; Fetal alloimmune thrombocytopenia
MeSH Terms: interventions — Immunoglobulins, Intravenous; Prednisone

STUDY DESIGN:
Intervention Model Description: randomization between 2 groups
Masking Description: participants and their physicians will know if they are receiving IVIG x 2 or IVIG x1 plus prednisone
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVIG x 2 (Experimental): IVIG 2 g/kg/wk divided into 2 infusions per week for women with a fetus affected by FNAIT
  Interventions: Drug: IVIG (Intravenous Immunoglobulin)
- IVIG x 1 + prednisone (Experimental): IVIG 1 g/kg/wk in 1 infusion per week + prednisone 0.5 mg po daily for women with a fetus affected by FNAIT
  Interventions: Drug: IVIG (Intravenous Immunoglobulin); Drug: prednisone

INTERVENTIONS:
Drug: IVIG (Intravenous Immunoglobulin) — one gram per kg of IVIG per infusion given either once or twice
Drug: prednisone — in arm with IVIG 1 gm/kg/wk will also receive prednisone 0.5 mg/kg/day
  Arms: IVIG x 1 + prednisone

SUMMARY:
The purposes of this study are to provide medical management by giving treatment to the mother that will bring up the fetal platelet count and to minimize the number of invasive procedures to the fetus (which may result in serious fetal injuries).

ELIGIBILITY:
Inclusion Criteria:

Pregnant women are eligible for inclusion into the Very High Risk Group if they:

* are PLA-1 (platelet antigen A1) negative and have known platelet incompatibility with their fetus
* have had a previous child who suffered an antenatal hemorrhage prior to 28 weeks gestation (as best as could be estimated)
* are less than 19 weeks gestation

Pregnant women are eligible for inclusion into the High Risk Group if they:

* are PLA-1 negative and have known platelet incompatibility with the fetus
* have had a previous child who suffered an antenatal hemorrhage after 28 weeks gestation (as best as could be estimated)
* are between 12-30 weeks gestation

Pregnant women are eligible for inclusion into the Standard Risk Group if they:

* are PLA-1 negative and have known platelet incompatibility with the fetus
* have not had a previous child who suffered an antenatal hemorrhage
* are between 20-30 weeks gestation

Exclusion Criteria:

Women are not eligible for inclusion into the Very High Risk Group if they:

* have had a previous child who suffered an antenatal hemorrhage after 28 weeks gestation
* are greater than 19 weeks gestation

Women are not eligible for inclusion into the High Risk Group if they:

* have had a previous child who suffered an antenatal hemorrhage prior to 28 weeks gestation
* are greater than 30 weeks gestation

Women are not eligible for inclusion into the Standard Risk Group if they:

* have had a previous child who suffered an antenatal hemorrhage
* are greater than 30 weeks gestation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2001-04; Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Bussel, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Cornell Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Lakkaraja M, Jin JC, Manotas KC, Vinograd CA, Ferd P, Gabor J, Wissert M, Berkowitz RL, McFarland JG, Bussel JB. Blood group A mothers are more likely to develop anemia during antenatal intravenous immunoglobulin treatment of fetal and neonatal alloimmune thrombocytopenia. Transfusion. 2016 Oct;56(10):2449-2454. doi: 10.1111/trf.13779. Epub 2016 Sep 9. PMID 27611703
- [Derived] Berkowitz RL, Lesser ML, McFarland JG, Wissert M, Primiani A, Hung C, Bussel JB. Antepartum treatment without early cordocentesis for standard-risk alloimmune thrombocytopenia: a randomized controlled trial. Obstet Gynecol. 2007 Aug;110(2 Pt 1):249-55. doi: 10.1097/01.AOG.0000270302.80336.dd. PMID 17666597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: pregnant women with a fetus affected by FNAIT were enrolled at multiple sites with local IRB permission and local consents fetuses were tracked in utero and after birth for 2 weeks
Groups:
- Intravenous Gammglobulin (IVIG) 1g/kg Twice Per Week: 51 women entered the study and received IVIG 1g/kg twice per week rounded off to the nearest 5-10 kg. The initial treatment weight was used throughout.
  premeds were diphenhydramine, acetaminophen and single dose prednisone as needed if the fetal platelet count was < 50,000/ul or not obtained at approximately 32 weeks of gestation either for technical reasons or parental refusal, prednisone 0.5mg/kg/day was added to the continued IVIG infusions delivery was primarily by Caesarean section unless the fetal count was known or strongly suspected to be (> 50,000 all women had fetal and neonatal alloimmune thrombocytopenia with a previous affected pregnancy and virtually all had parental incompatibility of HPA-1a ultrasound of the fetus was performed every 4 weeks or so and postnatally neonatal platelet counts were obtained and treatment of the fetus with platelet transfusion and/or IVIG and/or steroids was given as needed as determined by the NICU staff where the baby was delivered
- IVIG 1g/k/Week and Prednisone 0.5 mg/kg/Day: IVIG was infused at 1 gram/kg/week rounded off to the nearest 5-10 kg. The initial treatment weight was used throughout. premeds were diphenhydramine, acetaminophen and single dose prednisone as needed all women had fetal and neonatal alloimmune thrombocytopenia with a previous affected pregnancy and were known to be carrying an affected fetus treatment was initiated at approximately 20-26 weeks of gestation at approximately 32 weeks of gestation a fetal platelet count was obtained if the fetal platelet count was < 50,000/ul or was not obtained for either technical difficulty or patient refusal, then a second 1g/kg/week of IVIG was added until delivery delivery was typically by C/S unless the fetal platelet count was known or strongly suspected to be > 50,000/up neonatal platelet counts were obtained and treatment of the fetus with platelet transfusion and/or IVIG and/or steroids was given as needed as determined by the NICU staff where the baby was delivered
Period: Overall Study
Arm/Group | Intravenous Gammglobulin (IVIG) 1g/kg Twice Per Week | IVIG 1g/k/Week and Prednisone 0.5 mg/kg/Day
Started | 51 | 51
Completed | 51 | 48 (3 women chose to withdraw because they felt the study was "too inconvenient".)
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: study describes pregnant women who are receiving treatment but also fetuses and then newborns
Groups:
- IVIG (Intravenous Gamma Globulin) 2g/kg/Week: pregnant women with alloimmune thrombocytopenia and a previous affected fetus/newborn and a current affected fetus starting IVIG 2 g/kg/week
- IVIG 1g/kg/wk and Prednisone 0.5mg/kg/Day: pregnant women with alloimmune thrombocytopenia and a previous affected fetus/newborn and a current affected fetus starting IVIG 1 g/kg/week + prednisone 0.5mg/kg/day
- Total: Total of all reporting groups
Arm/Group | IVIG (Intravenous Gamma Globulin) 2g/kg/Week | IVIG 1g/kg/wk and Prednisone 0.5mg/kg/Day | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 102
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 102
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 46 | 94
  Canada | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Newborns With a Birth Platelet Count > 50,000/uL
Description: this uses the birth platelet count of the fetuses from the study when they are born
Time Frame: 32-40 weeks (the endpoint is the birth which is not at the same number of weeks for all of the babies. This is why the weeks are not listed specifically eg week 40
Measure: Number; unit: number of newborns with >50,000 pets
Groups:
- IVIG 1g/kg Twice Per Week: 51 women entered the study and received IVIG 1g/kg twice per week rounded off to the nearest 5-10 kg. The initial treatment weight was used throughout.
  premeds were diphenhydramine, acetaminophen and single dose prednisone as needed if the fetal platelet count was < 50,000/ul or not obtained at approximately 32 weeks of gestation either for technical reasons or parental refusal, prednisone 0.5mg/kg/day was added to the continued IVIG infusions delivery was primarily by Caesarean section unless the fetal count was known or strongly suspected to be (> 50,000 all women had fetal and neonatal alloimmune thrombocytopenia with a previous affected pregnancy and virtually all had parental incompatibility of HPA-1a ultrasound of the fetus was performed every 4 weeks or so and postnatally neonatal platelet counts were obtained and treatment of the fetus with platelet transfusion and/or IVIG and/or steroids was given as needed as determined by the NICU staff where the baby was delivered
Arm/Group | IVIG 1g/kg Twice Per Week | IVIG 1g/k/Week and Prednisone 0.5 mg/kg/Day
Number analyzed (Participants) | 51 | 51
number of newborns with >50,000 pets | 48 | 47

2. Secondary Outcome: Intracranial Hemorrhage: Number Occurring in Fetuses and Newborns of Mothers in Study
Description: number of ICH assessed by fetal and neonatal ultrasound with MRI back up most commonly in utero so range from 20-40 weeks fo gestation
Time Frame: time of ICH (range 20-40 wks)
Measure: Number; unit: number of newborns with ICH
Arm/Group | IVIG 1g/kg Twice Per Week | IVIG 1g/k/Week and Prednisone 0.5 mg/kg/Day
Number analyzed (Participants) | 51 | 51
number of newborns with ICH | 0 | 0

3. Secondary Outcome: Number of Fetal Platelet Counts > 50,000/uL
Description: Number of Fetal Platelet Counts > 50,000/uL Among Those Who Underwent Fetal Blood Sampling and Had a Fetal Platelet Count Determined
Time Frame: 32 +/- 2 weeks
Measure: Number; unit: number newborns with >50,000 pats
Arm/Group | IVIG 1g/kg Twice Per Week | IVIG 1g/k/Week and Prednisone 0.5 mg/kg/Day
Number analyzed (Participants) | 51 | 51
number newborns with >50,000 pats | 44 | 43

ADVERSE EVENTS:
Time Frame: collected for study women from 20 weeks of gestation until 2 weeks after birth of newborn fetus and newborns were collected for the same period of time
Groups:
- IVIG X 2 Weekly: Intravenous Immunoglobulin (IVIG) one gram per kg bodyweight infused twice weekly to mothers during pregnancy
  fetuses followed by serial ultrasound including after birth and newborns followed for 2 or so weeks after birth
- IVIG 1 g/kg/wk + Prednisone: intravenous gammaglobulin 1 g/kg/wk infused once weekly to mother and prednisone 0.5 mg/kg/day taken by mothers during pregnancy and then tapered after birth fo newborn
  fetuses followed by serial ultrasound including after birth and newborns followed for 2 or so weeks after birth
- IVIG X 2 Weekly--fetuses/Newborns: fetuses and newborns of mother receiving IVIG x 2 weekly
- IVIG x 1 + Prednisone---fetuses/Newborns: fetuses and newborns of mother receiving IVIG x 1 weekly + prednisone 0.5mg/kg daily
Arm/Group | IVIG X 2 Weekly | IVIG 1 g/kg/wk + Prednisone | IVIG X 2 Weekly--fetuses/Newborns | IVIG x 1 + Prednisone---fetuses/Newborns
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 14/51 | 12/51 | 4/51 | 3/51
Other Adverse Events (participants affected / at risk) | 12/51 | 8/51 | 0/51 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG X 2 Weekly (N=51) | IVIG 1 g/kg/wk + Prednisone (N=51) | IVIG X 2 Weekly--fetuses/Newborns (N=51) | IVIG x 1 + Prednisone---fetuses/Newborns (N=51)
preterm labor (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) — 1 aseptic meningitis
amnionitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gestational diabetes (Endocrine disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) — requiring hospitalization
HELLP (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — hypertension liver low platelets
thrombosis, venous (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Peripheral Intravenous Catheter thrombosis
depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
diabetes mellitus (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
fetal ICH (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Intracranial hemorrhage occurring in fetus
premature delivery (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3) | 4 (4) | 3 (3) — delivery prior to 35 weeks of gestation
neonatal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — sepsis in newborn
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG X 2 Weekly (N=51) | IVIG 1 g/kg/wk + Prednisone (N=51) | IVIG X 2 Weekly--fetuses/Newborns (N=51) | IVIG x 1 + Prednisone---fetuses/Newborns (N=51)
jaw tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — past history
IVIG dose error (Product Issues) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — once each: 10 grams and 120 grams
hypertension (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
bells palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
diabetes mellitus (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
neonatal hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — low blood sugar in newborn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No